CLINICAL TRIAL: NCT06973954
Title: Determination of Variables Associated With the Activation Level of Diabetic Individuals and Improvement of Activation Level
Brief Title: Improving the Activation Level of Diabetic Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülsüm Yıldız, Nurse, PhD Student, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Dokuz EU- HSE-IMN Phd- GY-01
Record Dates: First submitted 2025-04-19; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus (DM); Type 2 Diabetes Mellitus (T2DM); Patient Activation; Diabetes Self-management
Keywords: Diabetes Mellitus; Type 2 Diabetes Mellitus; Patient Activation; Patient Activation İnterventions; Improving Patient Activation
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Patient Participation

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled study planned in two stages: descriptive and experimental. In the first descriptive stage, variables related to the activation level of diabetic viruses were determined. Data were collected from 151 diabetic individuals. The second experimental planned stage was conducted on 30 individuals in the experimental group and 30 individuals in the control group, determined by randomization from 151 diabetic individuals whose data were collected in the first stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiment group (Message Sent) (Active Comparator): The experimental group consisted of 30 diabetic individuals. As an intervention, it was planned to send short messages containing information about diabetes, created by the researcher, to the diabetic individuals in the experimental group. The short messages were planned to be sent 3 days a week for 8 weeks.
  Interventions: Other: Text Message Intervention
- Control Group (Message not sent) (No Intervention): The control group consists of 30 diabetic individuals. No intervention will be applied to the control group.

INTERVENTIONS:
Other: Text Message Intervention — This intervention was prepared by the researcher with the support of artificial intelligence to increase the activation of diabetic individuals in the experimental group. It consists of short messages with the themes of gain, loss and motivation related to diabetes and self-management.
  Arms: Experiment group (Message Sent)

SUMMARY:
This study was planned to determine the activation levels of diabetic individuals and to improve the activation level. The study, planned as a descriptive and experimental type, is an attempt to increase the activation level of diabetic individuals.

DETAILED DESCRIPTION:
Type 2 diabetes, which is rapidly increasing in prevalence worldwide and poses a global threat, is a complex, chronic condition that requires ongoing medical care with multifactorial risk reduction strategies in addition to glucose management. 1 It causes serious physical and psychological distress to patients and their families, and also imposes a heavy economic burden on society. "2, 3, 4 Therefore, treatment of type 2 diabetes and prevention of its complications are particularly important. Self-management is the key to effective management and control of diabetes. 2, 5 Self-management, which includes activities such as diet, physical activity, self-monitoring of blood sugar, foot care, adherence to medication, and prevention of complications in managing symptoms and lifestyle changes associated with type 2 diabetes , is considered the cornerstone of diabetes management. "2, 6, 7, 8, 9, 10, 11" Individuals with chronic diseases such as type 2 diabetes need to participate in health care services to achieve better self-management and better health outcomes. The basis for this is patient activation. Patient activation refers to the knowledge, skills, and confidence of an individual in managing their own health and health care. Patient activation is the driving force of self-management. 12 Literature shows that individuals with high activation levels use more self-management services, exhibit better self-management behaviors such as diet, physical activity, and adherence to treatment plans, and tend to show optimal clinical outcomes such as HbA1c, high-density lipoproteins (HDL), blood pressure, and triglycerides. "2, 8, 12, 13, 14" In addition, more active adult patients believe they are in control of their own health. 17, 18 Highly activation patients show greater self-efficacy, higher quality of life, and lower depression scores. "17, 19, 21, 22, 23, 24, 25" Patients who demonstrate low levels of activation are often apathetic and depressed, have low health-related knowledge, low goal orientation, and poor compliance with any preventive health regimen or treatment, viewing their health as the responsibility of their physicians .

Positive health outcomes obtained with increased patient activation have led researchers to work on activating individuals. Studies examining the factors associated with activation in diabetic individuals are limited. Based on the data obtained from these studies, factors associated with patient activation have been grouped under three headings: demographic, clinical, and psychosocial factors. Demographic factors associated with patient activation have been reported in the literature as age, level of education, gender, race, marital status, and income status. In clinical factors, healthy nutrition, regular exercise, regular health screening, better diabetes control, body mass index, and positive health perception have been found to be associated with patient activation. Psychosocial factors associated with patient activation have been reported as health literacy, patient satisfaction, quality of life, level of hope, negative disease perception, self-efficacy, and depression.

Despite this evidence, there is insufficient literature on the determinants of patient activation in developing countries like ours. The aim of our study is to determine the variables associated with activation in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Having diabetes for 1 year or more, Able to read and write Turkish, Having no visual, auditory, perceptual or any other physical disability, Having the physical, mental and emotional capacity to participate in self-care activities, Having no language problems, Accepting to participate voluntarily in the study.

Exclusion Criteria:

* Individuals with any mental/cognitive problems,

  * Those who cannot read or write,
  * Those with visual, hearing, perception or any physical disability,
  * Those who are immobile or bedridden,
  * Those who do not have the ability to participate in their own self-care activities,
  * Those who do not want to participate in the study were excluded from the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure | 6 months
  In the first stage of our research, planned as descriptive, the following questions were sought.
  In this stage, the Patient Activation Level Measurement Tool (PAM), socio-demographic and disease-related characteristics questionnaire, and the Multidimensional Diabetes Questionnaire were used to measure the activation level of diabetic individuals.
  Are the socio-demographic characteristics of diabetic individuals related to the activation level? Are the disease-related characteristics of diabetic individuals related to the activation level? Are the perceived obstacles, perceived severity, perceived self-efficacy, perceived support, perceived outcome expectations of diabetic individuals evaluated with the multidimensional diabetes questionnaire related to the activation level?
Patient Activation Level | 6 months
  In the second experimental phase of the study, it is planned to increase the activation level of diabetic individuals with an intervention. The activation level of diabetic individuals is determined with the Patient Activation Level Measurement Tool (PAM). PAM is a valid, highly reliable, unidimensional, Guttman-type scale. It consists of 13 items. Activation is a four-stage process: 1. Believing in the importance of taking an active role, 2. Knowledge and confidence to take action, 3. Taking action, 4. Maintaining routine even under stress. Activation scores range from 0 to 100. Stage 1: lowest activation: 0-47, Stage 2: 47.1 - 55.1, Stage 3: 55.2 - 67.0, Stage 4: highest activation: 67.1-100 (Hibbard, et al, 2004).

SECONDARY OUTCOMES:
Self-care Behaviors, Metabolic Control Values, Self-Effectiveness Level | 6 months
  The difference between the self-care behaviors of individuals with diabetes participating in the program and those in the control group will be measured. Self-care behavior will be measured with the Diabetes Self-Care Scale. The Diabetes Self-Care Scale is a Likert-type scale and consists of 35 items. The self-care of patients who scored more than 66% of the scale was determined to be at an acceptable level. According to the 4-point Likert-type, the minimum acceptable level of the scale was determined as 92 points. The maximum score of the scale is 140, and as the score increases, the patients' ability to perform self-care activities increases positively. Self-Efficacy level was assessed with the "Self-Efficacy Scale for Type 2 Diabetics". A high score obtained from this Likert-type scale consisting of 20 items indicates a high level of self-efficacy. Metabolic values include fasting-postprandial blood sugar, HbAc, HDL, LDL, total cholesterol levels. Taken from routine measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Büyükkaya Besen, Associate professor, Study Director — Dokuz Eylul University Faculty of Nursing
Locations (1):
- Dokuz Eylul University Health Sciences Institute Izmir, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No